CLINICAL TRIAL: NCT01417442
Title: Association Of Prognosis And BRAF V600E Mutations In Papillary Thyroid Carcinoma
Brief Title: BRAF V600E Mutations In Papillary Thyroid Carcinoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Yeliz E. Ersoy, BEZMIALEM VAKIF UNIVERSITY
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011/5
Record Dates: First submitted 2011-07-06; First posted 2011-08-16 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-08

CONDITIONS: Papillary Thyroid Carcinoma
Keywords: papillary thyroid carcinoma; BRAF V600E; poor prognosis; aggressive
MeSH Terms: conditions — Thyroid Cancer, Papillary; Aggression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BRAF V600E POSITIVITY (Experimental): This mutation will be analysed using the tumor tissues of the patients operated for thyroid diseases and diagnosed with papillary thyroid carcinoma. And mutation positive patients will be investigated for the aggressive characteristics of the tumor.
  Interventions: Genetic: BRAF V600E POSITIVITY

INTERVENTIONS:
Genetic: BRAF V600E POSITIVITY — BRAF V600E mutation analysis will be made using the tumor tissues of the patients with papillary thyroid cancer (3 sections of 7 mm from he paraffin blocks). And mutation positives and negatives will be identified.

SUMMARY:
The purpose of this study is to determine whether BRAF V600E mutation in our patients with papillary thyroid cancer has an association with poor prognosis.

DETAILED DESCRIPTION:
Papillary thyroid carcinoma (PTC) is the most common type of thyroid malignancy and BRAF V600E mutation is the most common genetic alteration identified in PTC, ranging from 25 to 80%, with the average rate about 45%. Various studies demonstrated a relationship between BRAF V600E mutation and aggressive characteristics of the cancer, including the worse patient prognosis. But,there are no studies from Turkey regarding this topic. So the investigators will examine BRAF V600E mutation in our patients with PTC and try to assess the role of this mutation in prognosis and further management of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with papillary thyroid cancer

Exclusion Criteria:

* Patients who do not want to be a part of this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
BRAF V600E MUTATION | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Yeliz Emine Ersoy, Istanbul, Istanbul, Turkey (Türkiye)